CLINICAL TRIAL: NCT04811456
Title: MultiOrgan Inflammatory Syndromes COVID-19 Related Study
Acronym: MOIS-CoR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Wrocław Medical University (Unknown); University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: MOIS-CoR
Record Dates: First submitted 2021-03-22; First posted 2021-03-23 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: MIS-C; PIMS-TS; COVID-19; hyperinflammation; children
MeSH Terms: conditions — COVID-19; pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MIS-C: Cases fulfilling following criteria:
  1. fever ≥3 days
  2. at least two of the following:
     * rash or bilateral conjunctivitis or mucocutaneous inflammation signs
     * hypotension
     * features of myocardial dysfunction, pericarditis, or coronary artery abnormality, based on echocardiographic findings or elevated B-type natriuretic peptide (BNP)/N-terminal-pro-BNP (NT-proBNP) or troponin
     * evidence of coagulopathy
     * acute gastrointestinal problems
  3. elevated inflammatory markers AND
  4. no other apparent microbial cause
  5. evidence of COVID-19 (positive real-time polymerase chain reaction, antigen test or serology), or personal history of COVID-19 or contact with a proven COVID-19 case
  Interventions: Other: multisystem inflammatory syndrome in children (MIS-C)

INTERVENTIONS:
Other: multisystem inflammatory syndrome in children (MIS-C) — as in group description

SUMMARY:
The study comprise a nationwide, voluntary, on-line survey of inflammatory syndromes in children for retrospective (since 4th March 2020) and prospective data collection. Our aim was to capture and describe multisystem inflammatory syndrome in children (MIS-C) in Poland.

DETAILED DESCRIPTION:
The voluntary surveillance for retrospective (since 4th March) and prospective data collection was initiated under the National Consultant of Pediatrics auspices. Anonymized patient data from pediatric hospitals from all over the country are extracted from electronic and paper records and collected through online form developed for that purpose. Before the surveillance was launched, reporting clinicians underwent an online training, which included the current state of knowledge about multisystem inflammatory syndrome in children (MIS-C). Patient management is at the discretion of the relevant treating clinicians.

KD and aKD were defined following the American Heart Association (AHA) guidelines.

TSS was established based on modified criteria by the Centers for Disease Control and Prevention.

MAS was diagnosed based on the Paediatric Rheumatology International Trials Organization (PRINTO) criteria for MAS classification.

The definition of the inflammatory syndrome was based on the WHO MIS-C definition with the exclusion of SARS-CoV-2 confirmation.

For patients who met the inclusion criteria, demographic data, past medical history, data on COVID-19 exposure, clinical symptoms, physical examination findings, laboratory, imaging, and cardiologic tests results, treatment, and outcome data are collected.

All study definitions are defined in accordance to relevant guidelines and evaluated automatically with the use of a dedicated software.

ELIGIBILITY:
Inclusion Criteria:

* patients who required hospitalization since 4th March 2020;
* diagnosed Kawasaki disease (KD) or incomplete (atypical) Kawasaki disease (aKD) or toxic shock syndrome (TSS) or macrophage activation syndrome (MAS) or unspecified inflammatory syndrome;

Exclusion Criteria:

* other infectious and non-infectious causes that could be responsible for the disease

SARS-CoV-2 polymerase chain reaction (PCR) or serology result could have been positive or negative. Due to limited availability and reliability of serologic testing, proven or likely COVID-19 criterion was not a condition determining inclusion to the registry.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 0-18 years old hospitalized with inflammatory conditions
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
PICU | 5 years
  pediatric intensive care unit treatment need

SECONDARY OUTCOMES:
Heart dysfunction | 5 years
  Heart dysfunction is defined as ejection fraction (EF) of <55% and severe heart dysfunction as EF <35%.
CAA | 5 years
  Coronary artery abnormalities comprise both coronary dilation and/or coronary aneurysm. Dilation was defined by Z-score between 2 to 2.5, while aneurysm by Z score ≥2.5
Hypotension | 5 years
  Hypotension is defined by a minimal systolic blood pressure (sBP) below 70+2×age (in years) mmHg or below 90 mmHg for children >10 years old

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Okarska-Napierała, Principal Investigator — Medical University of Warsaw
Locations (2):
- Poland (2):
  - Medical University of Warsaw Children's Hospital, Warsaw
  - Wroclaw Medical University, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided